CLINICAL TRIAL: NCT04225936
Title: An Open-label, Two-Part, Single-dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BMS-986263 in Participants With Varying Degrees of Hepatic Impairment
Brief Title: A Single-dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BMS-986263 in Participants With Varying Degrees of Liver Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM025-015
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group A: Mild Hepatic Impairment (Experimental): Part 1
  Interventions: Drug: BMS-986263
- Group B: Moderate Hepatic Impairment (Experimental): Part 1
  Interventions: Drug: BMS-986263
- Group C: Severe Hepatic Impairment (Experimental): Part 2
  Interventions: Drug: BMS-986263
- Group D: Normal Hepatic function (control group) (Experimental): Part 1
  Interventions: Drug: BMS-986263
- Group E: Normal Hepatic Function (optional, control group) (Experimental): Part 2
  Interventions: Drug: BMS-986263

INTERVENTIONS:
Drug: BMS-986263 — Single Dose

SUMMARY:
The primary purpose of this study is to evaluate the effect of liver impairment on the safety and pharmacokinetics (PK) of BMS-986263

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* BMI ≥ 18 kg/m^2 and weight ≥ 50 kg at screening (BMI = weight [kg]/height [m^2]).
* Participants with normal hepatic function as judged by the investigator
* Participants with hepatic impairment as judged by the investigator

Exclusion Criteria:

* Clinically relevant abnormal medical history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests at screening that the investigator judges as likely to interfere with the objectives of the trial or the safety of the participant.
* Any major surgery within 4 weeks of study drug administration
* Previous exposure to BMS-986263

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) of components of BMS-986263 for injection | Day 1 to Day 31
Area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) of components of BMS-986263 for injection | Day 1 to Day 31
Area under the serum concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) of components of BMS-986263 for injection | Day 1 to Day 31
Total body clearance (CL) of components of BMS-986263 for injection | Day 1 to Day 31
Volume of distribution (Vz) of components of BMS-986263 for injection | Day 1 to Day 31
Terminal elimination half-life (T-Half) of components of BMS-986263 for injection | Day 1 to Day 31

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 31 days
Incidence of Serious Adverse Events (SAEs) | Up to 59 days or up to 30 days after dosing (whichever is longer)
Incidence of AEs leading to discontinuation | Nonserious AEs: Up to 31 days ; SAEs: Up to 59 days or up to 30 days after dosing (whichever is longer).
Number of participants with abnormalities in clinical laboratory assessments | Up to 59 days
Number of participants with vital sign abnormalities | Up to 59 days
Number of participants with 12-lead electrocardiogram (ECG) abnormalities | Up to 59 days
Number of participants with physical examination abnormalities | Up to 59 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- The Texas Liver Institute, San Antonio, Texas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm